CLINICAL TRIAL: NCT05911581
Title: Investigation of the Effect of Washing Solutions at Different Temperatures Used in Intra-arterial Cannulation for Invasive Blood Pressure Measurement by Doppler Ultrasonography
Brief Title: The Effect of the Use of Washing Solutions at Different Temperatures Used in Intra-arterial Cannulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Assoc.Phd.M.D, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/06-1
Record Dates: First submitted 2023-06-02; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Intrarterial Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- room temperature washing solution (Active Comparator): İntra-arterial flushing with heparinized fluid kept in room air
  Interventions: Other: intra-arterial flushing
- washing solution at patient temperature (Active Comparator): Intra-arterial flushing with heparinized fluid at patient body temperature
  Interventions: Other: intra-arterial flushing

INTERVENTIONS:
Other: intra-arterial flushing — The catheter will be flushed to prevent occlusion after radial artery catheterization.
  intra-arterial flushing with heparinized fluid kept in room air
  Other Names: group room
  Arms: room temperature washing solution
Other: intra-arterial flushing — Intra-arterial flushing with heparinized fluid at patient body temperature
  Other Names: group patient
  Arms: washing solution at patient temperature

SUMMARY:
Nowadays, intraarterial catheterization is frequently used as an invasive method for intraoperative blood pressure monitoring and control.The radial artery is frequently used in this procedure and the cannula should be flushed with 2-3 ml of heparinized fluid intermittently to prevent occlusion. During the operation, the ambient temperature is approximately 22-24 C and the patient temperature can be 34-36 C. Since the flushing fluids are also in the environment, they are 22-24 C. The aim of this study is to determine whether the fluids at room temperature cause vasoconstriction in the vessel and cause a change in blood pressure arterial values.

DETAILED DESCRIPTION:
The aim of this study is to determine whether room temperature fluids cause vasoconstriction or vasodilatation in the vessel and cause a change in blood pressure arterial values.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III risk class,
* Medically undergoing intra-arterial cannulation
* Being between the ages of 18-70

Exclusion Criteria:

* Diagnosis of DM
* Vascular disease,
* Bleeding diathesis,
* inotropic drug use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-16 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Arterial flow velocities PSV | 30th seconds after arterial flush
  After flushing performed , peak systolic velocity (PSV) values in the radial artery by Ultrasound doppler method.
Arterial flow velocities End-diastolic velocity | 30th seconds after arterial flush
  After flushing performed , end- diastolic velocity (EDV) values in the radial artery by ultrasound doppler method;
Arterial flow velocities resistive indices | 30th seconds after arterial flush
  After flushing performed resistive indices (RI) values in the radial artery by ultrasound doppler method.

SECONDARY OUTCOMES:
invasive and non-invasive blood pressure | 10th,30th,60th,90th ,120th and 150th seconds
  After flushing performed systolic, diastolic, and average blood pressure values measured

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No